CLINICAL TRIAL: NCT00119639
Title: A Study to Evaluate the Effect of Renal Function on the Single-Dose Pharmacokinetics of Sorafenib (BAY 43-9006, Nexavar).
Brief Title: Study to Evaluate the Effect of Renal Function on the Single-Dose Pharmacokinetics of BAY 43-9006
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11804
Record Dates: First submitted 2005-07-08; First posted 2005-07-14 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Kidney Diseases
MeSH Terms: conditions — Kidney Diseases | interventions — Sorafenib

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Sorafenib (BAY43-9006, Nexavar)

INTERVENTIONS:
Drug: Sorafenib (BAY43-9006, Nexavar) — All subjects were given a open-label, single dose of 400mg sorafenib

SUMMARY:
This is a 400 mg (2 x 200 mg tablets) sorafenib single dose, open-label study being conducted to compare the pharmacokinetics of plasma and urine and safety of sorafenib in subjects with severe, moderate, and mild renal impairment with those exhibiting normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal females
* Surgically sterile females
* Body Mass Index between 18-37
* Subjects with Clcr greater than 80 mL/min
* Subjects with Clcr 50 to 80 mL/min
* Subjects with Clcr 30 to 50 mL/min
* Clcr less than 30 mL/min but not on dialysis
* Subjects must test negative for HIV
* Subjects must test negative for drugs of abuse at screening

Exclusion Criteria:

All Subjects :

* Concomitant Medication: Treatment with CYP3A4 inducers, such as rifampin and St. John's Wort within 14 days of Day 1 until they leave the clinic on Day 7
* Donation of blood within 30 days of Day 1
* Recent participation in an investigational drug study during which active medication was given within 30 days of Day 1
* History of gastrointestinal disorder that could result in incomplete absorption of study drug
* Malignancy
* Significant neurologic or psychiatric disorders
* History of drug or alcohol abuse in year prior to screening for this trial, or current intake or >14 standard alcoholic drinks per week
* Prior history of epilepsy or other seizure disorders
* Known hypersensitivity to inhibitors of raf kinase or VEGFR-2
* Females of child-bearing potential
* Smoking > 10 cigarettes/day or equivalent
* Excessive consumption (more than five 8-oz. cups/day) of coffee or caffeine

Healthy Volunteer:

* Existing failure of a major organ system, or a medical disorder that would impair the subject's ability to complete the study (in the opinion of the investigator or the sponsor), eg history of blood coagulation disorders
* Hematocrit value < 34% in the control group at screening

Renal Impairment Groups:

* Existing failure of a major organ system or a medical disorder (other than the target disease) which would impair the subject's ability to complete the study (in the opinion of the investigator or the sponsor)
* Concomitant Medication: Renal impairment subjects taking phosphate binders, ion exchange resins and/or iron supplements may take them with their meals, but must withhold them on the morning of Day 1 (dosing day) until after their 4 hour post-dose tests and procedures are performed.
* Myocardial infarction, coronary artery bypass graft or percutaneous transluminal coronary angiography within 6 months of Day 1; unstable angina; uncontrolled significant hypertension within 3 months of Day 1; cerebral vascular accident or transient ischemic attack within 12 months of Day 1
* Subjects with hypertension who have had a medication or dose change within one week of Day 1
* Subjects requiring dialysis
* Subjects with kidney transplants
* Liver transaminase (AST, ALT) greater than 5 times the ULN at screening; any active liver disease or unexplained or persistent elevations in liver function tests
* Hematocrit value < 24% in the renal impaired groups

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-06; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of sorafenib in plasma and urine; single-dose safety of sorafenib in patients with renal impairment | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer